CLINICAL TRIAL: NCT07142772
Title: EMeRiT: Quantitative Assessment of the Etiologies of Megalencephaly Associated With a Detectable Tumor Risk
Brief Title: Quantitative Assessment of the Etiologies of Megalencephaly Associated With a Detectable Tumor Risk
Acronym: EMeRiT
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231309
Record Dates: First submitted 2025-04-23; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Megalocephaly
Keywords: Megalencephaly; tumor; Etiology
MeSH Terms: conditions — Megalencephaly; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children having macrocephaly with or without neurodevelopmental disorders: Children having macrocephaly ≥+3 SD due to brain MRI-confirmed MEG, with or without neurodevelopmental disorders, who have undergone genome sequencing

SUMMARY:
This study will show the value of early genetic diagnosis in the case of MEG in a child and may lead to recommendations aimed at preventing tumor risk based on a simple and easily accessible clinical criterion (the measurement of head circumference). Ultimately, this study may improve cancer prognosis in the population of children with MEG.

DETAILED DESCRIPTION:
During paediatric follow-up, head circumference (CP) measurement can detect severe macrocephaly (CP ≥ +3 SD) in 1% of the population, in individuals with or without neurodevelopmental disorder (NDD). After prescribing brain imaging showing excess brain growth or megalencephaly (MEG), pediatricians can refer patients to expert centers (Rare Disease Reference Centers) for an etiologic search for MEG. Genome sequencing is then prescribed by pediatric neurologists or geneticists as part of the "cerebral malformations" pre-indication (Plan France Genomic Medicine 2025).

In the literature, more than 70 genetic causes of MEG have been identified, 9 of which are responsible for pathologies associated with a sufficiently high tumor risk (>5%) to justify recommendations for regular screening, specific to each pathology ((Cowden, Simpson-Golabi-Behmel syndrome, Gorlin syndrome, neurofibromatosis type 1, variant in the DICER1 gene).

These genetic diseases are inconsistently associated with NDD (about 50%) and require specific follow-up to improve the oncological prognosis. The absence of an etiological diagnosis in these patients is potentially damaging and represents a theoretical loss of opportunity with regard to tumor risk. There are no large studies investigating the etiologies of MEGs, so the incidence of pathologies with tumor risk in this population remains unknown, with the exception of PTEN gene mutations, identified in 10% of patients with TND and MEG. This study will indicate the incidence of mutations in genes with tumor risk, which may eventually justify modifying current paediatric practice by recommending early etiological testing for MEGs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with macrocephaly ≥ +3 DS due to brain MRI-confirmed MEG with or without NDD
2. Patient with a proposal to investigate a genetic etiology by genome sequencing
3. No objection by the patient's parents or guardians
4. Patients affiliated to a social security scheme

Exclusion Criteria:

* Patients with an etiological diagnosis of its MEG
* Patients who have previously undergone genetic testing as part of their MEG, with or without a diagnosis
* Patients who have not received the standard-of-care genetic analysis, specifically whole genome sequencing

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Children having macrocephaly ≥+3 SD due to brain MRI-confirmed MEG, with or without neurodevelopmental disorders, who have undergone genome sequencing
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Characterization of the etiologies of MEGs associated with tumor risk in 200 children with or without NDD, who underwent genome sequencing. | Within 6 Months after last patient inclusion
  The investigator will study the diagnostic performance, i.e. the proportion in the sample of class 4 (probably pathogenic) or 5 (pathogenic) variants according to the American College of Medical Genetics (ACMG) classification

SECONDARY OUTCOMES:
To compare the diagnostic returns of the 2 patient groups | Within 6 Months after last patient inclusion
To establish a ranking of the yields of the 9 known MEG genes associated with tumor risk | Within 6 Months after last patient inclusion
  The investigator will do a descriptive analysis of the number of variants, their relative and absolute frequency.risk
To identify the nature and frequency of other genetic causes of MEG, apart from the 9 targeted genes | Within 6 Months after last patient inclusion
  The investigator will do a descriptive analysis of the number of variants, their relative and absolute frequency.risk
To establish genotype-phenotype correlations in the different etiologies found | Within 6 Months after last patient inclusion
  A descriptive analysis will be performed without statistical assumptions.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig HEIDE, medical doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- service Génétique clinique Pitié-Salpêtrière / Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No